CLINICAL TRIAL: NCT00897663
Title: Optimizing EGFR Inhibitor-Based Therapies for GBM
Brief Title: Improving the Selection of Patients With Glioblastoma Multiforme for Treatment With Epidermal Growth Factor Receptor Inhibitor Therapies
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: N0477; NCCTG-N0477; CDR0000527337 (Registry Identifier: PDQ (Physician Data Query)); NCI-2009-00645 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult gliosarcoma; adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Gene Expression Profiling; Microarray Analysis; Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group: Tissue samples from patients enrolled on clinical trials NCCTG-N0177 or NCCTG-N0074 are analyzed by microarray analysis and immunohistochemistry for biological markers predicting progression-free survival and overall survival. Biological markers include epidermal growth factor expression, vIII mutant p53 gene, P-AKT, p7056k, S6, 4EBP1, STAT-3, PLC-g, Erk, ErbB2, ErbB3, ErbB4, platelet-derived growth factor receptor, IGF1R, interleukin-6, FADD, and MGMT.
  Interventions: Genetic: gene expression analysis; Genetic: microarray analysis; Genetic: protein expression analysis; Other: diagnostic laboratory biomarker analysis; Other: immunohistochemistry staining method

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: protein expression analysis
Other: diagnostic laboratory biomarker analysis
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This laboratory study is looking at tissue samples from patients with glioblastoma multiforme to identify biomarkers that may improve the selection of patients for epidermal growth factor receptor inhibitor therapies.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify molecular characteristics that predict for overall survival and progression-free survival of patients treated with erlotinib hydrochloride, temozolomide, and radiotherapy on clinical trial NCCTG-N0177.

Secondary

* Identify molecular characteristics that predict for overall survival and progression-free survival of patients treated with gefitinib after radiotherapy on clinical trial NCCTG-N0074.

OUTLINE: This is a multicenter study.

Tissue samples from patients enrolled on clinical trials NCCTG-N0177 or NCCTG-N0074 are analyzed by microarray analysis and immunohistochemistry for biological markers predicting progression-free survival and overall survival. Biological markers include epidermal growth factor expression, vIII mutant p53 gene, P-AKT, p7056k, S6, 4EBP1, STAT-3, PLC-g, Erk, ErbB2, ErbB3, ErbB4, platelet-derived growth factor receptor, IGF1R, interleukin-6, FADD, and MGMT.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
All patients entered onto N0177 and N0074 who have appropriate archived clinical specimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tissue samples from patients enrolled on clinical trials NCCTG-N0177 or NCCTG-N0074.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Molecular characteristics that predict for overall survival and progression-free survival | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jann Sarkaria, MD, Study Chair — Mayo Clinic
Locations (10):
- United States (10):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota